CLINICAL TRIAL: NCT06705868
Title: Time-restricted Eating in Patients With Metabolic-associated Steatotic Liver Disease . CHRONOMASLD: A Chrononutrition/Chronotoxicity Randomized Controlled Trial.
Brief Title: Chrononutrition/ Chronotoxicity Intervention in People With Metabolic-associated Steatotic Liver Disease.
Acronym: CHRONOMASLD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus University of Technology (Other)
Collaborators: Cyprus State Heath Organization Services (Unknown)
Responsible Party: Principal Investigator, Konstantinos Makris, Professor of Environmental Health, Cyprus University of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHRONOMASLD
Record Dates: First submitted 2024-11-23; First posted 2024-11-26 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: MASLD; MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease; NAFLD; NAFLD - Non-Alcoholic Fatty Liver Disease; NAFLD (Nonalcoholic Fatty Liver Disease)
Keywords: non alcoholic fatty liver disease (NAFLD); chrononutrition; intermittent fasting; randomized controlled trial (RCT); chronotoxicity; time restricted eating; MASLD; Metabolic Dysfunction-Associated Steatotic Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Intermittent Fasting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Group A-Control) (Other): Participants in Group A will follow a Standard of Care Intervention. They will receive guidance on a) energy restriction, b) weight reduction, c) the macronutrient composition of the diet, d) limitation of alcohol intake (below the risk threshold of 30g/d and 20g/day for men and women, respectively) and e) increase their physical activity levels. Additionally, in this study patients will be asked to consume the general recommendation of "5-a-day" as part of their dietary healthier behaviour. Moreover, participants should stay well hydrated and get adequate of sleep (an average of 6 consecutive hours at night). Oral and written guidance for the management of MASLD will be administered. The duration of the intervention is 3 months.
  Interventions: Other: Lifestyle Management
- Time-restricted eating (Group B-Intervention) (Experimental): Participants will have to adhere to an ad libitum TRE dietary pattern (8 hours eating, 16 hours fasting) with an additional dietary restriction regarding the "5-a-day" fruit and vegetable in which they will need to be consumed between 9am-4pm. Some more restrictions regarding first and last meal will be asked. Participants will be instructed that their first meal of the day should not start for at least an hour after wake-up hour and will also be asked to have their last meal at least 2 hours earlier than bedtime (actual time of sleep). The duration of the intervention is 3 months.
  Interventions: Other: Diet-Time-restricted eating (TRE)

INTERVENTIONS:
Other: Diet-Time-restricted eating (TRE) — Ad libitum time-restricted scheme with a further time-restriction on fruit and vegetable consumption in participants with MASLD
  Arms: Time-restricted eating (Group B-Intervention)
Other: Lifestyle Management — The SoC intervention refers to an adaptation of a healthier lifestyle in elements that have to do with weight management, adopting healthier dietary habits, alcohol intake reduction, increase physical activity levels, in people diagnosed with MASLD.
  Arms: Standard of Care (Group A-Control)

SUMMARY:
The goal of this clinical trial is to study the effect of a time-restricted eating (TRE) dietary pattern combined with a time of consumption restriction about the daily portions of fruits and vegetables in people diagnosed with metabolic dysfunction-associated steatotic liver disease (MASLD).

The protocol of the study is an intention to treat protocol. The main research questions are:

1. Does compliance in a TRE dietary scheme (positively) affect changes in body weight and body fat mass in people diagnosed with MASLD?
2. Does an additional time restriction on the consumption of fruits and vegetables within the "light-window" of the day affects the metabolism of food contaminants?

Participants will be asked to:

1. Adhere to a TRE dietary pattern for 3 months. TRE consists of an 8-hour eating vs 16 hours fasting within the day. First meal of the day should not occur at least an hour after wake-up time and last meal of the day should occur not later than 2 hours before bed-time.
2. Adhere to a further time restricted consumption of a "5-a-day" portions of fruits and vegetables between the "light-window hours" between 9am to 4pm.
3. Visit the Nutrition & Dietetics Clinic once every month for anthropometric measurements (on 4 time points).
4. Collect and deliver first morning urine samples (on 7 time points).
5. Collect and deliver saliva samples at baseline and at the end of the trial (Saliva collection should occur every 4-hours for 48-hours including fasting collection at baseline and at the end of three months)

5) Complete a compliance and lifestyle questionnaire questionnaire via telephone interview to the research team every 2 weeks.

6) Share photos to the research team with the use of an application on time of actual fruit and vegetables consumption, 3-4 times per week throughout the study protocol.

Researchers will compare the designed intervention package of this TRE with the Standard of Care (SoC) protocol (based on the international guidelines) that is currently used in daily practice for the management of MASLD.

DETAILED DESCRIPTION:
This parallel-arm, randomized controlled trial (RCT) will study the effects of an ad libitum TRE dietary pattern (8 hours eating, 16 hours fasting) with an additional restriction regarding the fruit and vegetable consumption on health parameters, pesticide metabolism and concomitant toxicity in MASLD patients compared with the Standard of Care (SoC) approach, that will serve as the control group. Participants will be asked to consume all meals/snacks during the 8 hours daily period that they will select for themselves without any further dietary advice regarding caloric or other macronutrient intake. However, participants will be instructed that their first meal of the day should not start for at least an hour after wake-up hour and will also be asked to have their last meal at least 2 hours earlier than bedtime (actual time of sleep). Additionally, participants will have to consume 5 portions (400g) of fruits and vegetables within time-window for fruit & vegetable consumption earlier in the day; from 9am to 4pm.

Non-caloric beverage consumption (water, black coffee, unsweetened tea, non-sweetened beverages) will be allowed within the restricted hours of the intervention.

Participants allocated in the SoC group (control) will receive oral and written SoC lifestyle advice from a registered dietitian. The SoC advice is based on the EASL/EASD/EASO joint Clinical Practice Guidelines for the management of MASLD. Patients will receive guidance on a) energy restriction, b) weight reduction, c) the macronutrient composition of the diet, d) limitation of alcohol intake (below the risk threshold of 30g/d and 20g/day for men and women, respectively) and e) increase their physical activity levels. Additionally, in this study patients will be asked to consume standard "5-a-day" portions of fruits and vegetables daily, as part of their dietary healthier behaviour.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index 25 (±0,5)-45(±0,5) kg/m2
2. Clinical diagnosis of MASLD, not excluding undiagnosed NASH or with NASH stage F0-F1
3. Self-reported habitual eating period more than or equal to 14 h per day, BUT NOT LESS.
4. Cyprus inhabitants of for at least 1 year
5. Registered to the National Health System of the Republic of Cyprus (Gesy

Exclusion Criteria:

1. Night Shift worker
2. Fasting >12-h/day more than once a week or > once a week no food intake after 18:00
3. Co-existing causes of chronic liver disease according to standard diagnostic testing including, but not restricted to:

   1. Positive hepatitis B surface antigen
   2. Positive hepatitis C virus RNA
   3. Suspicion of drug-induced liver disease
   4. Alcoholic liver disease
   5. Autoimmune hepatitis
   6. Wilson's disease
   7. Hemochromatosis
   8. Primary biliary cholangitis or primary sclerosing cholangitis
   9. Known or suspected hepatocellular carcinoma
4. Medications which cause liver disease or secondary hepatic steatosis (Tamoxifen, systemic corticosteroids, methotrexate, tetracycline, estrogens, valproic acid, and statin (registration is possible if statin is delivered in a consistent dosage within 12 weeks)
5. Current or recent history (<5 years) of significant alcohol intake (>30g of alcohol/ day or >210g/week for men, >20g of alcohol/day or >140g/week for women)
6. Doctor diagnosed diabetes mellitus on insulin or sulfonylureas
7. Severe medical comorbidities [ischemic heart disease, 3rd degree atrioventricular block, chronic obstructive pulmonary disease, severe hypertension (blood pressure >200/120 mmHg)]
8. Unstable weight (>5% change in the last 2 months) or participation in a weight-loss program within the past 12 weeks
9. Sleep disorder (with a medical diagnosis) or individuals self-reporting sleep difficulties and poor sleep [average sleep less than 6 consecutive hours or patients who systematically experience sleep interruption for more than 2 times each night (waking up for toilet use is not to be considered sleep interruption)]
10. Individuals with food allergies (or hypersensitivity to the fruits and vegetables that will be selected for the study)
11. Systematic organic products consumers (defined as a self-reported usual consumption of more than 80% of their weekly fruits & vegetables being organic)
12. Pregnant or trying to become pregnant or lactating women
13. People not in position to communicate in Greek or English language
14. Having metallic parts in the body.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-12-15 (Estimated); Study Completion 2029-12-15 (Estimated)

PRIMARY OUTCOMES:
Changes in body weight | From enrolment to the end of treatment at 3 months (with two in-between measurement)
  Changes in body weight (in kilograms) from baseline to the end of intervention in the TRE and the Soc group (intervention vs control, respectively). Depending on the data distribution, independent samples t-test or Wilcoxon Rank-Sum Test will be used If the changes do or do not follow a normal distribution between baseline and post-treatment are normally distributed, respectively. Mixed Effect Models will be used to assess the main and interaction (included if p<0.05) effects between groups and time since study initiation adjusting for confounders, including circadian rhythm metrics such as melatonin and/or cortisol.
Changes in body fat mass | From enrolment to the end of treatment at 3 months (with one in-between measurement)
  Changes in body fat mass (expressed as % of the total body weight in kilograms) from baseline to the end of intervention in the TRE and the Soc group (intervention vs control, respectively). Depending on the data distribution, independent samples t-test or Wilcoxon Rank-Sum Test will be used If the changes do or do not follow a normal distribution between baseline and post-treatment are normally distributed, respectively. Mixed Effect Models will be used to assess the main and interaction (included only if p<0.05) effects between groups and time since study initiation adjusting for confounders, including circadian rhythm metrics such as melatonin and/or cortisol.

SECONDARY OUTCOMES:
Changes in Pesticide Metabolite 3-phenoxybenzoic Acid (3-PBA) Levels in Urine | From first day of the intervention to the end of treatment at 3 months (with six in between measurements)
  Change in Pesticide Metabolite 3-phenoxybenzoic Acid (3-PBA) Levels in Urine (in µg/L, corrected for creatinine levels) between the TRE and the SoC intervention. Percent change in pesticide metabolite 3-phenoxybenzoic acid (3-PBA) levels between the last sample of the TRE group (intervention period) and the last sample of the SoC treatment period. The results of the linear-mixed effect models are the ones considered as they take into account the repeated measures for each participant and the TRE treatment duration adjusting for confounders, including circadian rhythm metrics such as melatonin and/or cortisol.
Changes in Pesticide Metabolite 6-chloronicotininc Acid (6-CN) Levels in Urine | From first day of the intervention to the end of treatment at 3 months (with six in between measurements)
  Change in Pesticide Metabolite 6-chloronicotininc Acid (6-CN) Levels in Urine (in µg/L, corrected for creatinine levels) between the TRE and the SoC intervention. Percent change in pesticide metabolite 6-chloronicotininc Acid (6-CN) levels between the last sample of the TRE group (intervention period) and the last sample of the SoC treatment period. The results of the linear-mixed effect models are the ones considered as they take into account the repeated measures for each participant and the TRE treatment duration adjusting for confounders, including circadian rhythm metrics such as melatonin and/or cortisol.
Changes in waist circumference (WC) | From enrolment to the end of treatment at 3 months (with one in-between measurement)
  Changes in waist circumference (in centimetres) from baseline to the end of intervention in the TRE and the Soc group (intervention vs control, respectively). Depending on the data distribution, independent samples t-test or Wilcoxon Rank-Sum Test will be used If the changes do or do not follow a normal distribution between baseline and post-treatment are normally distributed, respectively. Mixed Effect Models will be used to assess the main and interaction (included if p<0.05) effects between groups and time since study initiation adjusting for confounders, including circadian rhythm metrics such as melatonin and/or cortisol.
Changes in 4-Hydroxynonenal (4HNE) Levels in Urine | From first day of the intervention to the end of treatment at 3 months (with six in between measurements)
  Change in Urine levels of the biomarker of oxidative stress 4-Hydroxynonenal (4HNE) (in µg/L, corrected for creatinine levels), between the TRE and the SoC intervention. Percent change in metabolite of oxidative stress of 4-Hydroxynonenal (4HNE) levels between the last sample of the TRE group (intervention period) and the last sample of the SoC treatment period. The results of the linear-mixed effect models are the ones considered as they take into account the repeated measures for each participant and the TRE treatment duration adjusting for confounders, including circadian rhythm metrics such as melatonin and/or cortisol.
Changes in Body Mass Index (BMI) | From enrolment to the end of treatment at 3 months (with two in-between measurement)
  Changes in Body Mass Index (in kilograms divided by meters in square) from baseline to the end of intervention in the TRE and the Soc group (intervention vs control, respectively). Depending on the data distribution, independent samples t-test or Wilcoxon Rank-Sum Test will be used If the changes do or do not follow a normal distribution between baseline and post-treatment are normally distributed, respectively. Mixed Effect Models will be used to assess the main and interaction (included if p<0.05) effects between groups and time since study initiation adjusting for confounders, including circadian rhythm metrics such as melatonin and/or cortisol.
Changes in glucose (Gluc) levels in blood | From enrolment to the end of treatment at 3 months (one measurement at the beginning and one measurement at the end of the intervention)
  Changes on blood's glucose (Gluc) levels (in mg/dL) from baseline to the end of intervention in the TRE and the Soc group (intervention vs control, respectively). Depending on the data distribution, independent samples t-test or Wilcoxon Rank-Sum Test will be used If the changes do or do not follow a normal distribution between baseline and post-treatment are normally distributed, respectively. Mixed Effect Models will be used to assess the main and interaction (included if p<0.05) effects between groups and time since study initiation adjusting for confounders, including circadian rhythm metrics such as melatonin and/or cortisol.
Changes in total cholesterol (TC) levels in blood | From enrolment to the end of treatment at 3 months (one measurement at the beginning and one measurement at the end of the intervention)
  Changes on blood's total cholesterol (TC) levels (in mg/dL) from baseline to the end of intervention in the TRE and the Soc group (intervention vs control, respectively). Depending on the data distribution, independent samples t-test or Wilcoxon Rank-Sum Test will be used If the changes do or do not follow a normal distribution between baseline and post-treatment are normally distributed, respectively. Mixed Effect Models will be used to assess the main and interaction (included if p<0.05) effects between groups and time since study initiation adjusting for confounders, including circadian rhythm metrics such as melatonin and/or cortisol.
Changes in high-density lipoprotein cholesterol (HDL) levels in blood | From enrolment to the end of treatment at 3 months (one measurement at the beginning and one measurement at the end of the intervention)
  Changes on blood's high-density lipoprotein cholesterol (HDL) levels (in mg/dL) from baseline to the end of intervention in the TRE and the Soc group (intervention vs control, respectively). Depending on the data distribution, independent samples t-test or Wilcoxon Rank-Sum Test will be used If the changes do or do not follow a normal distribution between baseline and post-treatment are normally distributed, respectively. Mixed Effect Models will be used to assess the main and interaction (included if p<0.05) effects between groups and time since study initiation adjusting for confounders, including circadian rhythm metrics such as melatonin and/or cortisol.
Changes in low-density lipoprotein cholesterol (LDL) levels n blood | From enrolment to the end of treatment at 3 months (one measurement at the beginning and one measurement at the end of the intervention)
  Changes on blood's low-density lipoprotein cholesterol (LDL) levels (in mg/dL) from baseline to the end of intervention in the TRE and the Soc group (intervention vs control, respectively). Depending on the data distribution, independent samples t-test or Wilcoxon Rank-Sum Test will be used If the changes do or do not follow a normal distribution between baseline and post-treatment are normally distributed, respectively. Mixed Effect Models will be used to assess the main and interaction (included if p<0.05) effects between groups and time since study initiation adjusting for confounders, including circadian rhythm metrics such as melatonin and/or cortisol.
Changes in alanine transaminase (ALT) levels n blood | From enrolment to the end of treatment at 3 months (one measurement at the beginning and one measurement at the end of the intervention)
  Changes on blood's alanine transaminase (ALT) levels (in U/IL) from baseline to the end of intervention in the TRE and the Soc group (intervention vs control, respectively). Depending on the data distribution, independent samples t-test or Wilcoxon Rank-Sum Test will be used If the changes do or do not follow a normal distribution between baseline and post-treatment are normally distributed, respectively. Mixed Effect Models will be used to assess the main and interaction (included if p<0.05) effects between groups and time since study initiation adjusting for confounders, including circadian rhythm metrics such as melatonin and/or cortisol.
Changes in aspartate aminotransferase (AST) levels in blood | From enrolment to the end of treatment at 3 months (one measurement at the beginning and one measurement at the end of the intervention)
  Changes on blood's aspartate aminotransferase (AST) levels (in U/IL) from baseline to the end of intervention in the TRE and the Soc group (intervention vs control, respectively). Depending on the data distribution, independent samples t-test or Wilcoxon Rank-Sum Test will be used If the changes do or do not follow a normal distribution between baseline and post-treatment are normally distributed, respectively. Mixed Effect Models will be used to assess the main and interaction (included if p<0.05) effects between groups and time since study initiation adjusting for confounders, including circadian rhythm metrics such as melatonin and/or cortisol.
Changes in C-Reactive Protein (CRP) levels n blood | From enrolment to the end of treatment at 3 months (one measurement at the beginning and one measurement at the end of the intervention)
  Changes on blood's C-Reactive Protein (CRP) levels (in mg/dL) from baseline to the end of intervention in the TRE and the Soc group (intervention vs control, respectively). Depending on the data distribution, independent samples t-test or Wilcoxon Rank-Sum Test will be used If the changes do or do not follow a normal distribution between baseline and post-treatment are normally distributed, respectively. Mixed Effect Models will be used to assess the main and interaction (included if p<0.05) effects between groups and time since study initiation adjusting for confounders, including circadian rhythm metrics such as melatonin and/or cortisol.

OTHER OUTCOMES:
Changes in other pesticide biomarkers in urine | From first day o the intervention to the end of treatment at 3 months (with six in between measurements)
  Change in Change in other pesticide biomarkers in Urine (in µg/L, corrected for creatinine levels) between the TRE and the SoC intervention. Percent change in any other measured pesticide metabolite between the last sample of the TRE group (intervention period) and the last sample of the SoC treatment period. The results of the linear-mixed effect models are the ones considered as they take into account the repeated measures for each participant and the TRE treatment duration. Levels in Urine (in µg/L, corrected for creatinine levels) between the TRE and the SoC intervention. Percent change in other pesticide biomarker levels between the last sample of the TRE group (intervention period) and the last sample of the SoC treatment period. The results of the linear-mixed effect models are the ones considered as they take into account the repeated measures for each participant and the TRE treatment duration, adjusting for confounders, including circadian rhythm metrics.
Changes in other biomarkers of oxidative stress in urine | From first day o the intervention to the end of treatment at 3 months (with six in between measurements)
  Change in other biomarkers of oxidative stress in Urine (in µg/L, corrected for creatinine levels) between the TRE and the SoC intervention. Percent change in any other measured biomarkers of oxidative stress between the last sample of the TRE group (intervention period) and the last sample of the SoC treatment period. The results of the linear-mixed effect models are the ones considered as they take into account the repeated measures for each participant and the TRE treatment duration. Levels in Urine (in µg/L, corrected for creatinine levels) between the TRE and the SoC intervention. Percent change in other pesticide biomarker levels between the last sample of the TRE group (intervention period) and the last sample of the SoC treatment period. The results of the linear-mixed effect models are the ones considered as they take into account the repeated measures for each participant and the TRE treatment duration adjusting for confounders, including circadian rhythm metrics.
Changes in metabolome in saliva and urine | From first day o the intervention to the end of treatment at 3 months (with six in between measurements)
  Change in metabolome profile in the 24-h in saliva or urine (in µg/L, corrected for creatinine levels) between the TRE and the SoC intervention. Percent change in metabolome profile between the last day samples of the TRE group (intervention period) and the last day samples of the SoC treatment period will be compared with an Exposome wide association analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Limassol General Hospital, Limassol, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided